CLINICAL TRIAL: NCT06077331
Title: A Multi-Center, Randomized, Double Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Efficacy and Safety of HS-10374 in Adult Subjects With Moderate To Severe Plaque Psoriasis
Brief Title: A Study to Evaluate Efficacy and Safety of HS-10374 for Moderate to Severe Plaque Psoriasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10374-201
Record Dates: First submitted 2023-08-24; First posted 2023-10-11 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HS-10374 Dose 1 (Experimental)
  Interventions: Drug: HS-10374 tablets 1mg; Drug: HS-10374 tablets 5mg; Drug: HS-10374-matched placebo tablets
- HS-10374 Dose 2 (Experimental)
  Interventions: Drug: HS-10374 tablets 1mg; Drug: HS-10374 tablets 5mg
- Placebo (Active Comparator)
  Interventions: Drug: HS-10374-matched placebo tablets

INTERVENTIONS:
Drug: HS-10374 tablets 1mg — Administered orally QD for 12 weeks
  Arms: HS-10374 Dose 1; HS-10374 Dose 2
Drug: HS-10374 tablets 5mg — Administered orally QD for 12 weeks
  Arms: HS-10374 Dose 1; HS-10374 Dose 2
Drug: HS-10374-matched placebo tablets — Administered orally QD for 12 weeks
  Arms: HS-10374 Dose 1; Placebo

SUMMARY:
This study has been designed to explore the clinical efficacy and safety of HS-10374 in the treatment of moderate to severe plaque psoriasis. Additionally, this study is to find the optimal dosing for the future clinical development of HS-10374.

DETAILED DESCRIPTION:
This is a 12-week, multi-center, randomized, double blind, placebo-controlled, Phase 2 study. The study duration includes a 4-week screening period, a 12-week treatment period, and a 4-week follow-up period. All eligible subjects will be randomly assigned to 1 of 3 treatment arms (HS-10374 Dose 1, HS-10374 Dose 2, and placebo) in an equal ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 18-70 years
2. Diagnosis of plaque psoriasis for at least 6 months
3. Eligible for phototherapy or systemic therapy
4. Plaque covering ≥ 10% of BSA
5. PASI ≥ 12, sPGA ≥3

Exclusion Criteria:

1. Diagnosis of non-plaque psoriasis or drug-induced psoriasis
2. Recent history of infection, history or risk of serious infection
3. Any major illness or evidence of unstable condition of major organ systems including psychiatric disease
4. Any condition possibly affecting the PK process of the study drug
5. Evidence of other skin conditions that would interfere with the evaluation of psoriasis
6. History of hypersensitivity to the ingredients of study drugs, history of anaphylaxis
7. History of lack of response to any therapeutic agent targeted to IL-12, IL-17 or IL-23 at approved doses after at least 3 months of therapy
8. Have received the prohibited treatment during the protocol required washout period
9. Any significant laboratory or procedure abnormalities that might place the subject at unacceptable risk during this study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with moderate to severe plaque psoriasis achieving PASI 75 response at Week 12 | Baseline to Week 12
  Psoriasis Area and Severity Index (PASI) is a scoring system quantifying the severity of psoriasis based on both lesion severity and area of involvement. PASI assessment is performed by investigators, and the numeric score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 75 response is defined as 75% or greater improvement in PASI score from baseline.

SECONDARY OUTCOMES:
Incidence, severity and association with the study drug of adverse events (AEs), serious AEs (SAEs), and AEs leading to discontinuation | Baseline to Week 16
Number of participants with clinical laboratory abnormalities | Baseline to Week 16
  Clinical laboratory tests include hematology, coagulation testing, blood chemistry, urinalysis, stool analysis, high-sensitivity C-reactive protein, etc.
Number of participants with abnormalities of vital signs | Baseline to Week 16
  Vital signs measured include blood pressure, pulse rate, and temperature.
Number of participants with abnormalities of physical examination | Baseline to Week 16
  Physical examination includes assessments of general appearance, skin, lymph nodes, head, neck, lung, heart, abdomen, spine, extremities, nervous system, etc.
Incidence of clinically significant changes in electrocardiogram (ECG) | Baseline to Week 16
  ECG parameters include heart rate, PR interval, RR interval, QRS duration, QTcF interval.
Proportion of patients with sPGA 0/1 at specified time points | Baseline to Week 16
  Static physician's global assessment (sPGA) of psoriasis is an average assessment of all psoriatic lesions based on erythema, induration, and scale. It's a 5-point scale performed by investigators. A sPGA score of 0 or 1 means "clear" or "almost clear" respectively.
PASI 50 response rates at specified time points | Baseline to Week 16
  Psoriasis Area and Severity Index (PASI) is a scoring system quantifying the severity of psoriasis based on both lesion severity and area of involvement. PASI assessment is performed by investigators, and the numeric score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 50 response is defined as 50% or greater improvement in PASI score from baseline.
PASI 75 response rates at specified time points | Baseline to Week 16
  Psoriasis Area and Severity Index (PASI) is a scoring system quantifying the severity of psoriasis based on both lesion severity and area of involvement. PASI assessment is performed by investigators, and the numeric score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 75 response is defined as 75% or greater improvement in PASI score from baseline.
PASI 90 response rates at specified time points | Baseline to Week 16
  Psoriasis Area and Severity Index (PASI) is a scoring system quantifying the severity of psoriasis based on both lesion severity and area of involvement. PASI assessment is performed by investigators, and the numeric score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 90 response is defined as 90% or greater improvement in PASI score from baseline.
PASI 100 response rates at specified time points | Baseline to Week 16
  Psoriasis Area and Severity Index (PASI) is a scoring system quantifying the severity of psoriasis based on both lesion severity and area of involvement. PASI assessment is performed by investigators, and the numeric score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 100 response is defined as 100% improvement in PASI score from baseline.
Change from baseline in PASI scores at specified time points | Baseline to Week 16
  Psoriasis Area and Severity Index (PASI) is a scoring system quantifying the severity of psoriasis based on both lesion severity and area of involvement. PASI assessment is performed by investigators, and the numeric score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity.
Change from baseline in BSA at specified time points | Baseline to Week 16
  Psoriasis body surface area (BSA) involvement is measured using the handprint method with the size of a patient's handprint representing ~1% of body surface area involved.
Change from baseline in DLQI scores at specified time points | Baseline to Week 16
  The dermatology life quality index (DLQI) is a patient reported outcome measurement. It's a questionnaire consisting of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week. Each question is scored on a scale of 0 to 3, and the sum of each scores range from 0 (no impairment of life quality) to 30 (maximum impairment).
Ctrough | Baseline to Week 12
  Trough observed plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Xu, Principal Investigator — Huashan Hospital; Yangfeng Ding, Principal Investigator — Shanghai Dermatology Hospital; Chao Ci, Principal Investigator — First Affiliated Hospital of Wannan Medical College; Weili Pan, Principal Investigator — Zhejiang Provincial People's Hospital; Shiqin Tao, Principal Investigator — Wuxi No. 2 People's Hospital; Yayu Hu, Principal Investigator — Taizhou University Affiliated Municipal Hospital; Tianhong Xu, Principal Investigator — The Third People's Hospital of Hangzhou; Zhu Shen, Principal Investigator — Guangdong Provincial People's Hospital; Mingkai Ji, Principal Investigator — The Second Affiliated Hospital of Xiamen Medical College; Chao Ji, Principal Investigator — First Affiliated Hospital of Fujian Medical University; Qing Guo, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Xiaohua Wang, Principal Investigator — Dermatology Hospital of Southern Medical University; Xiaoyong Zhou, Principal Investigator — Wuhan First Hospital; Zudong Meng, Principal Investigator — Shiyan City People's Hospital; Fengming Hu, Principal Investigator — Jiangxi Dermatology Hospital; Rong Xiao, Principal Investigator — The Second Xiangya Hospital, Central South University; Yu Wang, Principal Investigator — Affiliated Hospital of Guizhou Medical University; Tiechi Lei, Principal Investigator — Wuhan University People's Hospital; Yanyan Feng, Principal Investigator — Chengdu Second people's hospital; Rixin Chen, Principal Investigator — Nanyang city first People's Hospital; Chunshui Yu, Principal Investigator — Suining Central Hospital; Xiaojing Kang, Principal Investigator — Xinjiang Autonomous Region People's Hospital; Aijun Chen, Principal Investigator — First Affiliated Hospital of Chongqing Medical University; Jianguo Li, Principal Investigator — Henan Provincial People's Hospital; Yan Zhou, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Songmei Geng, Principal Investigator — The Second Affiliated Hospital of Xi 'an Jiaotong University; Guoqiang Zhang, Principal Investigator — The First Hospital of Hebei Medical University; Xinsuo Duan, Principal Investigator — The Affiliated Hospital of Chengde Medical College; Linfeng li, Principal Investigator — Beijing Friendship Hospital; Chunlei Zhang, Principal Investigator — Peking University Third Hospital; Shifa Zhang, Principal Investigator — North East Central International Hospital Limited; Shanshan Li, Principal Investigator — The First Hospital of Jilin University; Yuzhen Li, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University; Xiaodong Sun, Principal Investigator — Shenyang Hospital of Integrated Chinese and Western Medicine; Xinghua Gao, Principal Investigator — First Hospital of China Medical University
Locations (1):
- Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality, China